CLINICAL TRIAL: NCT07404410
Title: Robotic Technologies for APATHy in Dementia: a Randomised Controlled Trial (RAPHAel)
Acronym: RAPHAel
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Giovanna Zamboni (Other)
Collaborators: University of Genova (Other); Fondazione Don Carlo Gnocchi Onlus (Other); University of Florence (Other)
Responsible Party: Sponsor-Investigator, Giovanna Zamboni, Full Professor of Neurology | Department of Biomedical, Metabolic and Neural Sciences | University of Modena and Reggio Emilia; Consultant Neurologist | AOU Modena, University of Modena and Reggio Emilia
Organization: University of Modena and Reggio Emilia (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 263/2024/DISP/AOUMO
Record Dates: First submitted 2026-02-04; First posted 2026-02-11 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Apathy; Apathy in Dementia
Keywords: dementia; apathy; robotics
MeSH Terms: conditions — Lethargy; Dementia | interventions — Occupational Therapy; Standard of Care

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- telepresence robot (Experimental): The first experimental intervention uses a telepresence robotic system operated remotely by a trained researcher or therapist. Through this system, participants receive structured and personalized cognitive stimulation sessions delivered at home. The intervention protocol is based on evidence-supported cognitive rehabilitation programs and includes multiple weekly sessions over a six-week period. The telepresence robot enables real-time audiovisual interaction while allowing the operator to navigate the home environment, supporting engagement and continuity of care.
  Interventions: Behavioral: Occupational Therapy
- social robot (Experimental): The second experimental intervention involves a social humanoid robot deployed in the participant's home. The robot is connected to a dedicated conversational server that enables personalized verbal and non-verbal interactions. The system adapts conversations to the participant's interests, personal history, and interaction patterns. Interactions may be initiated by the participant or proactively by the robot, with the aim of stimulating conversational initiative, social engagement, and sustained attention. The frequency and duration of interactions are flexible within the predefined intervention period, allowing the intervention to integrate into daily routines.
  Interventions: Device: Pepper robot connected to a CAIR server
- occupational therapy (Active Comparator): The active control intervention consists of a structured home-based occupational therapy program targeting behavioral symptoms. This intervention focuses on meaningful activities, environmental adaptations, caregiver education, and strategies to support participation and motivation in daily life. The occupational therapy protocol reflects current standards of care and is delivered over the same six-week timeframe as the experimental interventions.
  Interventions: Device: telepresence robotic system

INTERVENTIONS:
Device: telepresence robotic system — The telepresence robot is designed to enable high-quality remote interaction through high-definition video streaming, clear two-way audio, and intuitive mobile navigation. It allows a therapist to connect in real time with a participant at home, moving within the environment and interacting as if physically present. In the RAPHAEL study, the telerobot is used by an occupational therapist to deliver personalized home-based sessions, guiding participants through exercises and activities via video calls conducted from the therapist's own device. The robot operates according to the manufacturer's intended use and user manual. Its modular hardware and software, reliability, and ease of use support consistent delivery of intervention sessions. The telerobot is already widely used in healthcare, education, and professional settings in more than 30 countries, making it a well-established platform for remote clinical interaction and support.
  Other Names: telerobot
  Arms: occupational therapy
Device: Pepper robot connected to a CAIR server — The intervention is based on an integrated robotic system designed to support personalized social interaction at home. It includes a commercial humanoid robot (Pepper) used as a physical interaction platform, supported by a local computer server and a Wi-Fi router with 4G connectivity to ensure stable operation. The core of the intervention is a dedicated software medical device (Server CAIR), which manages and adapts the interaction logic. A client application running on the robot enables verbal and non-verbal communication with the participant, while a separate software interface allows researchers to personalize content based on individual preferences and history. Speech recognition and language processing are supported by third-party services for voice transcription and response generation. Together, these components enable adaptive, conversational interactions aimed at stimulating engagement and social participation in a home setting.
  Other Names: social robot; talking robot; culturally sensitive robot
  Arms: social robot
Behavioral: Occupational Therapy — Human-based intervention delivered through an occupational therapy program focused on the prevention and management of behavioral symptoms, conducted by an occupational therapist in accordance with Essential Levels of Care (LEA). The techniques and protocols aim to prevent, reduce, and manage BPSD, train the caregiver, and improve quality of life for both the individual and the caregiver. The intervention includes 8 home visits and 2 telephone sessions over 6 weeks.
  Other Names: OT; standard of care
  Arms: telepresence robot

SUMMARY:
The goal of this trial is to learn whether home-based robotic interventions can reduce apathy in people with cognitive decline. Apathy means reduced motivation, interest, or initiative in daily life. It is a common and distressing symptom in people with mild cognitive impairment (MCI) or dementia and can strongly affect both participants and their caregivers.

This study will compare two different robotic interventions with standard occupational therapy. Researchers want to understand if these new technologies can help people become more engaged, motivated, and involved in everyday activities, and whether they also reduce stress and improve quality of life for caregivers.

The main questions this study aims to answer are:

* Do robotic interventions reduce apathy more than standard occupational therapy?
* Are these robotic interventions easy to use and acceptable for people with cognitive impairment?
* Do these interventions reduce caregiver stress and improve caregiver quality of life?

Participants will be adults over 40 years of age with a diagnosis of mild cognitive impairment or dementia caused by a neurodegenerative disease, such as Alzheimer's disease, frontotemporal dementia, or dementia with Lewy bodies. All participants must show clinically relevant apathy and have a family member or caregiver who can support them during the study and answer questionnaires.

Participants will be randomly assigned to one of three groups:

* A telepresence robot group, where participants interact at home with a therapist through a remotely controlled robot that delivers personalized cognitive stimulation.
* A social robot group, where participants interact at home with a humanoid robot that holds personalized conversations on topics of interest.
* A control group receiving home-based occupational therapy, which is the current standard care for behavioral symptoms.

Each intervention lasts six weeks and takes place in the participant's home. The robotic interventions are designed to fit into daily routines and can be adapted to the participant's abilities and preferences. Occupational therapy sessions focus on meaningful activities, environmental adaptations, and caregiver support.

Participants will complete assessments at three time points: before the intervention, at the end of the six-week intervention, and eight weeks after the intervention ends. These assessments include interviews, questionnaires, and simple tasks to measure apathy, emotional responses, social interaction, and quality of life. Caregivers will also complete questionnaires about stress and daily burden.

Researchers will also collect information about how often and how participants interact with the robots, such as how long conversations last and how engaged participants appear. These data will help researchers understand how robotic interactions relate to changes in apathy and behavior.

This study aims to provide evidence on whether robotic technologies can be safely and effectively used at home to support people with cognitive impairment and apathy. The results may help develop new non-drug treatments and improve care options for people living with dementia and their caregivers.

DETAILED DESCRIPTION:
Apathy is one of the most common behavioral symptoms associated with neurodegenerative disorders, including mild cognitive impairment (MCI) and dementia. It is characterized by diminished motivation, reduced initiation of activities, emotional blunting, and decreased social engagement. Apathy is associated with faster functional decline, reduced quality of life, increased caregiver burden, and limited response to currently available pharmacological treatments. For these reasons, non-pharmacological interventions are considered a priority target for clinical research.

This randomized controlled trial investigates the effectiveness of two home-based robotic interventions compared with standard occupational therapy for the management of apathy in individuals with cognitive decline. The study is conducted within a multi-center academic and clinical framework and follows international standards for interventional research, including SPIRIT recommendations and Good Clinical Practice principles.

The study adopts a single-blind, three-arm randomized design. Participants are randomly assigned in a 1:1:1 ratio to one of two experimental robot-based interventions or to an active control intervention consisting of home-based occupational therapy. Outcome assessments are performed by evaluators who are blinded to treatment allocation, while participants and intervention providers are aware of the assigned intervention due to the nature of the study.

The first experimental intervention uses a telepresence robotic system operated remotely by a trained researcher or therapist. Through this system, participants receive structured and personalized cognitive stimulation sessions delivered at home. The intervention protocol is based on evidence-supported cognitive rehabilitation programs and includes multiple weekly sessions over a six-week period. The telepresence robot enables real-time audiovisual interaction while allowing the operator to navigate the home environment, supporting engagement and continuity of care.

The second experimental intervention involves a social humanoid robot deployed in the participant's home. The robot is connected to a dedicated conversational server that enables personalized verbal and non-verbal interactions. The system adapts conversations to the participant's interests, personal history, and interaction patterns. Interactions may be initiated by the participant or proactively by the robot, with the aim of stimulating conversational initiative, social engagement, and sustained attention. The frequency and duration of interactions are flexible within the predefined intervention period, allowing the intervention to integrate into daily routines.

The active control intervention consists of a structured home-based occupational therapy program targeting behavioral symptoms. This intervention focuses on meaningful activities, environmental adaptations, caregiver education, and strategies to support participation and motivation in daily life. The occupational therapy protocol reflects current standards of care and is delivered over the same six-week timeframe as the experimental interventions.

All interventions are conducted in the participant's home environment to maximize ecological validity and generalization of effects. Where needed, technical support such as internet connectivity is provided to ensure consistent delivery of robot-based interventions. Participants and caregivers receive instruction on the use of devices, and safety procedures are implemented throughout the intervention period.

Assessments are conducted at baseline, immediately after the six-week intervention, and at follow-up six weeks after the end of treatment. These assessments include standardized clinical scales, behavioral tasks, and caregiver-reported measures. In addition, sensor-based and interaction-derived data are collected during selected tasks and robot interactions to explore digital markers of apathy and engagement. These data include measures related to movement kinematics, interaction frequency, conversational dynamics, and system usability.

Data are pseudonymized and stored in a secure electronic data capture system accessible only to authorized research personnel. Each participating center acts as an independent data controller for data collected locally, while centralized data management supports harmonization and analysis. All data handling procedures comply with applicable data protection regulations.

The primary aim of the study is to determine whether robotic interventions provide added value over standard occupational therapy in reducing apathy in people with cognitive impairment. Secondary aims include evaluating usability, feasibility, caregiver-related outcomes, and the relationship between clinical measures and digitally derived behavioral indicators.

By combining clinical assessments with advanced robotic technologies, this study seeks to generate evidence on innovative, scalable, and home-based approaches to the management of apathy. The findings are expected to inform future clinical practice and support the development of digital and robotic solutions for non-pharmacological treatment in neurodegenerative conditions.

ELIGIBILITY:
Inclusion Criteria:

* Age 40 years or older
* Clinical diagnosis of a neurocognitive disorder, including: Mild cognitive impairment (MCI) or mild behavioral impairment (MBI), or Major neurocognitive disorder (dementia), due to Alzheimer's disease, frontotemporal dementia, dementia with Lewy bodies, or other neurodegenerative diseases.
* Presence of clinically relevant apathy, defined as a score greater than 2 on the apathy domain (G) of the Neuropsychiatric Inventory (NPI).
* Preserved ability to understand and produce spoken and written language sufficient to participate in the intervention and assessments.
* Absence of clinically significant agitation or aggressiveness, defined as a score lower than 2 on the agitation/aggression domain (C) of the NPI.
* Adequate educational and occupational history sufficient to exclude intellectual disability.
* Availability of a study partner (family member, friend, or caregiver) who: Knows the participant well, Has contact with the participant for at least 10 hours per week, Is able to complete questionnaires about the participant, Is able to read, understand, and speak Italian, and Provides independent informed consent for participation.
* Ability and willingness of the participant (and study partner, when applicable) to provide informed consent.

Exclusion criteria:

* Refusal or withdrawal of informed consent by the participant or the study partner.
* History or current evidence of neurological conditions other than the target neurodegenerative diseases that may affect cognitive function (e.g., major stroke, brain tumor, normal pressure hydrocephalus, traumatic brain injury).
* History or current diagnosis of major psychiatric disorders that could interfere with study participation or assessments.
* Presence of medical conditions that may significantly affect cognitive function (e.g., severe renal or hepatic failure, untreated obstructive sleep apnea, hypothyroidism, vitamin B12 deficiency).
* Clinically significant agitation or aggressiveness, defined as a score of 2 or higher on the agitation/aggression domain (C) of the Neuropsychiatric Inventory (NPI).
* Inability to understand or communicate in Italian sufficient to complete study procedures.
* Absence of an eligible study partner or withdrawal of consent by the study partner.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2026-02-16 (Estimated); Primary Completion 2026-10-30 (Estimated); Study Completion 2026-11-30 (Estimated)

PRIMARY OUTCOMES:
Change in apathy severity | Baseline to 6 weeks
  Change in apathy severity measured by the Apathy Evaluation Scale (AES) total score, assessed from baseline (T0) to end of intervention at 6 weeks (T1).

SECONDARY OUTCOMES:
Caregiver burden | Baseline, 6 weeks
  Change in caregiver burden measured by the Zarit Burden Inventory (ZBI) total score.
caregiver quality of life | Baseline, 6 weeks
  Change in caregiver quality of life measured by the Quality of Life-Alzheimer's Disease (QoL-AD) caregiver version
social cognition | 0 to 6 weeks
  Change in social cognition performance measured by the Yoni-48 task and the Edinburgh Social Cognition Test (ESCoT).

IPD SHARING:
Plan to Share IPD: Undecided